CLINICAL TRIAL: NCT00755170
Title: A Phase II Study of the Combination of Metronomic Vinorelbine and Bevacizumab as 2nd Line Treatment in Patients With Non Small Cell Lung Cancer (NSCLC)
Brief Title: Metronomic Vinorelbine and Bevacizumab in Patients With Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.18
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Vinorelbine; Bevacizumab; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vinorelbine metronomic + bevacizumab
  Interventions: Drug: Vinorelbine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Vinorelbine — Metronomic vinorelbine (p.o) 30 mg total dose/day, every Monday, Wednesday and Friday of each week, continuously without intervals for the equivalence of 6 cycles maximum
  Other Names: Navelbine
Drug: Bevacizumab — Bevacizumab (IV) 10 mgr/Kgr on day 1 and 15 every 4 weeks for 6 cycles maximum followed by Bevacizumab (IV) 10 mgr/Kgr on day 1 and 15 every 4 weeks until disease progression
  Other Names: Avastin

SUMMARY:
This trial will evaluate the efficacy and safety of metronomic vinorelbine and bevacizumab combination in patients with pretreated, advanced non small cell lung cancer

DETAILED DESCRIPTION:
Intravenous (IV) vinorelbine is a standard chemotherapy option for the treatment of metastatic NSCLC, either alone or in combination with other agents such as CDDP or Carboplatin with overall response rates (ORR) of 15-35% as 1st line treatment and less than 10% as salvage treatment. For the past few years vinorelbine is available for per os (po) administration with acceptable and reliable pharmacokinetic profiles and with a bioavailability of approximately 40% of the IV dose. In randomized phase II studies IV and po vinorelbine have shown comparable response and overall survival rates. The low dose metronomic chemotherapy that is administered in short intervals has been shown in vitro an in vivo to have antiangiogenic effects. Bevacizumab is a well known anti-angiogenic agent. Recently, a phase III study of 1st line treatment in patients with advanced or metastatic NSCLC showed that the addition of bevacizumab to a platinum-based regimen provided a survival benefit. This study will evaluate the combination of metronomic vinorelbine and bevavizumab as 2nd line treatment of NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, metastatic (stage IV) non small cell lung cancer
* One previous platinum based chemotherapy regimen with or without taxanes for metastatic NSCLC
* Measurable disease, defined as at least 1 bidimensionally measurable lesion ≥ 20 X 10 mm
* Age ≥ 18 years
* Performance status (WHO) 0-2
* Life expectancy of at least 12 weeks
* Adequate bone marrow (ANC ≥ 1,500/mm3, PLT ≥ 100,000/mm3, Hgb ≥ 11 g/dL), liver (Bilirubin ≤ 1.5 upper normal limit, SGOT/SGPT ≤ 2.5 upper normal limit in the absence of liver metastases or ≤ 5 upper normal limit in the presence of liver metastases), and renal function (Creatinine ≤ 1,5 upper normal limit)
* Patients must be able to understand the nature of this study
* Written informed consent

Exclusion Criteria:

* Second primary malignancy, except for non-melanoma skin cancer. Pregnant or lactating women
* Any serious, uncontrolled comorbidity on the investigator's judgment
* Uncontrolled infection
* Any sustained chronic toxicity > grade 2 according to the NCI CTCAE (version 3.0)
* Brain metastases, except if radiated and asymptomatic
* Radiotherapy within the previous 4 weeks
* Previous radiotherapy to the only measurable lesion
* Proteinuria ≥ 500 mgr of protein daily
* Hemoptysis > 10 cc per event
* Clinically significant hematemesis
* Centrally located lesion or in contact with major vessels
* Pulmonary lesion with cavitation
* Documented hemorrhagic diathesis or coagulation disorder
* Cardiovascular disease (class II-IV NYHA congestive heart failure, myocardial infarction within the previous 4 months, unstable angina, LVEF < normal, ventricular arrhythmia, uncontrolled hypertension)
* Thrombotic event within the previous 6 months
* Concurrent use of aspirin > 325 mgr daily, low molecular weight heparin in therapeutic dose, warfarin or acenocoumarol, non-steroid anti-inflammatory agents
* Concurrent treatment with other anti-cancer drug
* Major surgical procedure within the previous 4 weeks
* Serum Να+ < 120mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Response rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment on each cycle
Progression free survival | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Agelaki, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki
  - Interbalkan Hospital, division of Oncology, Pylaia, Thessaloniki, Thessaloniki